CLINICAL TRIAL: NCT05042661
Title: National Taipei University of Nursing and Health Sciences
Brief Title: Acupuncture-like Transcutaneous Electrical Nerve Stimulation on Bowel Symptom and Quality of Life in Patients With Irritable Bowel Syndrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The number of cases accepted has reached expectations.
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Tsu Ying Fang, Principal investigator, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TFang
Record Dates: First submitted 2021-09-04; First posted 2021-09-13 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2023-02

CONDITIONS: Acupuncture-like Transcutaneous Electrical Nerve Stimulation; Irritable Bowel Syndrome
Keywords: irritable bowel syndrome; acupuncture-like transcutaneous electrical nervestimulation; quality of life
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupuncture-like transcutaneous electrical nerve stimulation (Experimental): 1. The experimental group received acupuncture-like transcutaneous electrical nerve stimulation three times a week for 4 weeks.
  2. Invention and control groups are 4 weeks and 3 weeks respectively. Each time will be for 20 minutes acupuncture-like transcutaneous electrical nerve stimulation treatment
  Interventions: Device: acupuncture-like transcutaneous electrical nerve stimulation
- Control group:conventional therapy (No Intervention): The control group will receive routine care.

INTERVENTIONS:
Device: acupuncture-like transcutaneous electrical nerve stimulation — The intervention group performed Al-TENS therapy 3 times a week for at least 20 minutes each time for 4 consecutive weeks. The second, fourth, and eighth week after the intervention.
  Arms: acupuncture-like transcutaneous electrical nerve stimulation

SUMMARY:
To discuss the effects of improving the irritable bowel syndrome patients' quality of life and defecation after implementing acupuncture-like Transcutaneous Electrical nerve stimulation.

DETAILED DESCRIPTION:
This experiment will use a clinical design that will collect cases in a local teaching hospital. The way of convenience sampling will gather from the irritable bowel syndrome patients. After a questionnaire, randomly to make invention and control groups. Invention and control groups are 4 weeks and 3 weeks respectively. Each time will be for 20 minutes acupuncture-like transcutaneous electrical nerve stimulation treatment. The Control group will still have normal nursing. There will be 72 patients in two groups. The measured timing will be in the second, fourth, and eighth weeks after the prediction and invention.

ELIGIBILITY:
Inclusion Criteria:

1. Those who are at least 20 years old (inclusive) and are willing to sign a written informed consent after explaining the purpose of the research.
2. A patient with irritable bowel syndrome diagnosed by a doctor for at least 6 months (inclusive).
3. Communicate in Mandarin or Hokkien.

Exclusion Criteria:

1. Those who cannot take care of themselves in daily life.
2. Those who have had severe abdominal and colorectal surgery.
3. Those who have been diagnosed with inflammatory bowel disease or colorectal cancer.
4. Those with a history of mental illness, such as schizophrenia and obsessive- compulsive disorder.
5. Women who are pregnant, breastfeeding, and less than 12 months after delivery.
6. Other serious diseases, such as acute myocardial infarction, endocrine disease, decompensated cirrhosis, stroke, and end-stage renal disease, etc.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-02-13 (Actual)

PRIMARY OUTCOMES:
WHOQOL-BREF,Taiwan version | pretest
  There are a total of 28 questions on this scale, of which 26 are common questions around the world, and the other 2 are local questions. This questionnaire is a positive question and a five-point scoring system. The higher the score, the better the quality of life.
WHOQOL-BREF,Taiwan version | 2 weeks after the pretest
  There are a total of 28 questions on this scale, of which 26 are common questions around the world, and the other 2 are local questions. This questionnaire is a positive question and a five-point scoring system. The higher the score, the better the quality of life
WHOQOL-BREF,Taiwan version | 4 weeks after the pretest
  There are a total of 28 questions on this scale, of which 26 are common questions around the world, and the other 2 are local questions. This questionnaire is a positive question and a five-point scoring system. The higher the score, the better the quality of life
WHOQOL-BREF,Taiwan version | 8 weeks after the pretest
  There are a total of 28 questions on this scale, of which 26 are common questions around the world, and the other 2 are local questions. This questionnaire is a positive question and a five-point scoring system. The higher the score, the better the quality of life
irritable bowel syndrome Severity Score | pretest
  There are a total of 5 questions on this scale. This questionnaire is a positive question type. The score of each item can be from 0 to 100. Therefore, the overall severity of IBS ranges from 0 to 500. The severity of symptoms can be divided into mild; moderate; severe, the higher the score, the more severe the IBS symptoms
irritable bowel syndrome Severity Score | 2 weeks after the pretest
  There are a total of 5 questions on this scale. This questionnaire is a positive question type. The score of each item can be from 0 to 100. Therefore, the overall severity of IBS ranges from 0 to 500. The severity of symptoms can be divided into mild; moderate; severe, the higher the score, the more severe the IBS symptoms
irritable bowel syndrome Severity Score | 4 weeks after the pretest
  There are a total of 5 questions on this scale. This questionnaire is a positive question type. The score of each item can be from 0 to 100. Therefore, the overall severity of IBS ranges from 0 to 500. The severity of symptoms can be divided into mild; moderate; severe, the higher the score, the more severe the IBS symptoms
irritable bowel syndrome Severity Score | 8 weeks after the pretest
  There are a total of 5 questions on this scale. This questionnaire is a positive question type. The score of each item can be from 0 to 100. Therefore, the overall severity of IBS ranges from 0 to 500. The severity of symptoms can be divided into mild; moderate; severe, the higher the score, the more severe the IBS symptoms
Irritable Bowel Syndrome Quality of Life | pretest
  This questionnaire has a total of 34 questions, all of which are positive questions, and are scored with five points, divided into 1 point = completely no, 2 points = a little bit, 3 points = medium, 4 points = equivalent, 5 points = extreme. The score range is 34~170 points, the higher the score, the worse the quality of life
Irritable Bowel Syndrome Quality of Life | 2 weeks after the pretest
  This questionnaire has a total of 34 questions, all of which are positive questions, and are scored with five points, divided into 1 point = completely no, 2 points = a little bit, 3 points = medium, 4 points = equivalent, 5 points = extreme. The score range is 34~170 points, the higher the score, the worse the quality of life
Irritable Bowel Syndrome Quality of Life | 4 weeks after the pretest
  This questionnaire has a total of 34 questions, all of which are positive questions, and are scored with five points, divided into 1 point = completely no, 2 points = a little bit, 3 points = medium, 4 points = equivalent, 5 points = extreme. The score range is 34~170 points, the higher the score, the worse the quality of life
Irritable Bowel Syndrome Quality of Life | 8 weeks after the pretest
  This questionnaire has a total of 34 questions, all of which are positive questions, and are scored with five points, divided into 1 point = completely no, 2 points = a little bit, 3 points = medium, 4 points = equivalent, 5 points = extreme. The score range is 34~170 points, the higher the score, the worse the quality of life
Bristol Stool Form Scale | pretest
  The first and second types of stool show that the patient has constipation, the first type is more serious than the second type; the normal stool types are the third and fourth types, and the fifth to seventh types are suspected Diarrhea (Lewis, & Heaton, 1997), the above description indicates that the lower the score, the more severe the constipation symptoms, and vice versa, the more severe the diarrhea symptoms
Bristol Stool Form Scale | 2 weeks after the pretest
  The first and second types of stool show that the patient has constipation, the first type is more serious than the second type; the normal stool types are the third and fourth types, and the fifth to seventh types are suspected Diarrhea (Lewis, & Heaton, 1997), the above description indicates that the lower the score, the more severe the constipation symptoms, and vice versa, the more severe the diarrhea symptoms
Bristol Stool Form Scale | 4 weeks after the pretest
  The first and second types of stool show that the patient has constipation, the first type is more serious than the second type; the normal stool types are the third and fourth types, and the fifth to seventh types are suspected Diarrhea (Lewis, & Heaton, 1997), the above description indicates that the lower the score, the more severe the constipation symptoms, and vice versa, the more severe the diarrhea symptoms
Bristol Stool Form Scale | 8 weeks after the pretest
  The first and second types of stool show that the patient has constipation, the first type is more serious than the second type; the normal stool types are the third and fourth types, and the fifth to seventh types are suspected Diarrhea (Lewis, & Heaton, 1997), the above description indicates that the lower the score, the more severe the constipation symptoms, and vice versa, the more severe the diarrhea symptoms

OTHER OUTCOMES:
Part 1: Basic personal information:Basic and disease information list 1 | pretest
  gender
Part 1: Basic personal information:Basic and disease information list 2 | pretest
  Date of birth
Part 1: Basic personal information:Basic and disease information list 3 | pretest
  marital status
Part 1: Basic personal information:Basic and disease information list 4 | pretest
  education level
Part 1: Basic personal information:Basic and disease information list 5 | pretest
  Work
Part 1: Basic personal information:Basic and disease information list 6 | pretest
  religion
Part 1: Basic personal information:Basic and disease information list 7 | pretest
  family history
Part 1: Basic personal information:Basic and disease information list 8 | pretest
  History of chronic disease
Basic and disease information list 9 | pretest
  smokes
Part 1: Basic personal information:Basic and disease information list 10 | pretest
  drink wine
Part 1: Basic personal information:Basic and disease information list 11 | pretest
  Betel nut
Part 1: Basic personal information:Basic and disease information list 12 | pretest
  Sleep status
Part 1: Basic personal information:Basic and disease information list 13 | pretest
  Special eating habits
Part 1: Basic personal information:Basic and disease information list 14 | pretest
  Exercise habits
Part 2: Symptoms of Irritable Bowel Syndrome:Basic and disease information list 1 | pretest
  Irritable bowel disease onset time
Part 2: Symptoms of Irritable Bowel Syndrome:Basic and disease information list 2 | pretest
  Bowel movement
Part 2: Symptoms of Irritable Bowel Syndrome:Basic and disease information list 3 | pretest
  treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Tsu Ying Fang, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided